CLINICAL TRIAL: NCT01284010
Title: Genome-Wide Analysis of Genetic Alterations in Adult Acute Lymphoblastic Leukemia
Brief Title: Biomarkers in Blood and Bone Marrow Samples From Patients With Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-21001; CALGB-21001; RC1CA145707 (NIH); P30CA014236 (NIH); CDR0000694150 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — In Situ Hybridization, Fluorescence; Gene Expression Profiling; Microarray Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Diagnostic, complete remission, and germ-line specimens are analyzed for DNA profiling and gene resequencing by the Affymetrix SNP6.0 microarray platform, PCR, and fluorescence in situ hybridization (FISH). Frequency of genetic alterations are performed by the Agilent 2100 Bioanalyzer. Results are then compared with the data already generated from pediatric patients.
  Interventions: Genetic: DNA analysis; Genetic: fluorescence in situ hybridization; Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: mutation analysis; Genetic: polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: fluorescence in situ hybridization
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in blood and bone marrow samples from patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To perform high-resolution, genome-wide profiling of DNA copy number alterations and loss-of-heterozygosity in samples from adult patients with acute lymphoblastic leukemia (ALL) obtained at diagnosis.
* To perform candidate gene resequencing of diagnostic ALL samples.
* To examine correlation of genetic alterations with outcome.
* To examine the correlation between microarray multi-gene and multi-exon expression signatures with specific alterations and outcome.
* To understand genetic events that contribute to the formation, development, and relapse of adult ALL by integrating the copy number and sequence alterations with the multi-gene signatures, and by comparing these data with data already generated in pediatric ALL.

OUTLINE: Diagnostic, complete remission, and germ-line specimens are analyzed for DNA profiling and gene resequencing by the Affymetrix SNP6.0 microarray platform, PCR, and fluorescence in situ hybridization (FISH). Frequency of genetic alterations are performed by the Agilent 2100 Bioanalyzer. Results are then compared with the data already generated from pediatric patients.

ELIGIBILITY:
Inclusion:

• Diagnostic and germ-line specimens from patients with acute lymphoblastic leukemia (ALL) treated on protocols CALGB 9511, CALGB-19802, CALGB-10001, CALGB-10102, and CALGB-10403 and who have been registered on the companion study CALGB-9665 (The CALGB Leukemia Tissue Bank)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute lymphoblastic leukemia (ALL) patients treated on protocols CALGB 9511, 19802, 10001, 10102, and 10403, and who have been registered on the companion study CALGB 9665 (The CALGB Leukemia Tissue Bank)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
complete remission rate | Up to 7 Years
disease free survival | Up to 7 Years
cumulative incidence of relapse | Up to 7 years
overall survival | Up to 7 years
event-free survival | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: James Downing, MD, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States